CLINICAL TRIAL: NCT02570126
Title: Safety and Immunogenicity Study of 2 Formulations of GSK Biologicals' Varicella Vaccines Given as a 2-dose Course in the Second Year of Life.
Brief Title: A Safety and Immune Study of 2 Types of GlaxoSmithKline's Varicella Vaccines Given as a 2-doses Course to Healthy Children 12-23 Months of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200147; 2013-003535-30 (EudraCT Number)
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Chicken-pox Illness (Varicella Virus Disease); Chickenpox
Keywords: Immunogenicity; Varicella; Safety; Human serum albumin; Healthy children; 12 to 23 months
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- VAR_HSA_F Group (Experimental): 2 doses of Varilrix HSA-free vaccine, one at Visit 1 (Day 0) and the other at Visit 2 (Day 42), will be given to the subjects in this group. The vaccine will be administered subcutaneously in the triceps region of the left arm
  Interventions: Biological: Varilrix HSA-free
- VAR Group (Active Comparator): 2 doses of Varilrix™ vaccine, one at Visit 1 (Day 0) and the other at Visit 2 (Day 42), will be given to the subjects in this group. The vaccine will be administered subcutaneously in the triceps region of the left arm
  Interventions: Biological: Varilrix™

INTERVENTIONS:
Biological: Varilrix HSA-free — 2 doses will be administered, one at Day 0 and the other at Day 42
  Arms: VAR_HSA_F Group
Biological: Varilrix™ — 2 doses will be administered, one at Day 0 and the other at Day 42
  Arms: VAR Group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of 2 formulations of GSK Biologicals' varicella vaccines given as a 2-dose course in the second year of life.

DETAILED DESCRIPTION:
GSK Biologicals has removed human serum albumin (a stabilizer) from its varicella vaccine to minimize as much as possible the use of animal or human-derived products in the production of vaccines. The study is intended to provide information on the safety and immunogenicity of GlaxoSmithKline (GSK) Biologicals' candidate varicella vaccine formulated without human serum albumin (HSA) in contrast to Varilrix™ (GSK) which contains HSA when both are used in a two-dose schedule, with the first and second doses given approximately 42 days apart in the second year of life.

The immunogenicity sub-cohort will be comprised of approximately 400 subjects, representing approximately 100 subjects enrolled in each of the participating countries.

Rationale for amendment 1: Sites in the UK can perform home visits. For subjects participating through home visits, the subject's parent(s) / Legally Acceptable Representative(s) [LAR(s)] will be requested to sign a Recruitment/Randomisation agreement to provide personal information and to agree to have their child randomised before providing written consent to participate in the study (to be provided at the 1st home visit).

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/ LAR(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 23 months of age (i.e. 12 months to a day before 24 months) at the time of the first study vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* Subjects in stable health as determined by investigator's clinical examination and assessment of subject's medical history.
* Subjects must have had prior administration of a dose of measles, mumps and rubella (MMR) vaccine at least 30 days (Day -31 or earlier) prior to study vaccination at Day 0.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the day of study vaccination (i.e., 30 days prior to Visit 1/Day 0) or planned use during the entire study period.
* Concurrently participating in another clinical study, in which the child has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration (defined as 14 or more consecutive days) of immunosuppressants, or other immune-modifying drugs during the period starting 180 days prior to the first vaccine dose or any planned administration of immunosuppressive and immune-modifying drugs during the entire study.

  * For corticosteroids, this will mean prednisone ≥0.5 mg/kg/day or equivalent.
  * Inhaled and topical steroids are allowed.
* Planned administration/ administration of a live viral vaccine not foreseen by the study protocol during the period starting 30 days prior to study vaccination at Visit 1/Day 0 until study end. Non study live viral vaccines can be administered at Visit 3 (Day 84) after completion of study procedures.
* Planned administration/ administration of an inactivated vaccine not foreseen by the study protocol during the period starting 7 days prior to each vaccination (at Visit 1/Day 0 and Visit 2/Day 42) and ending 14 days after each vaccination. Outside of this period, non-study inactivated vaccines can be administered as per standard of care.
* Administration of immunoglobulins and/or any blood products during the period starting 180 days prior to the first vaccine dose or planned administration from the date of first study vaccination through the entire study.
* History of varicella or zoster.
* Known exposure to varicella/zoster during the period starting within 30 days prior to first study vaccination.
* Previous vaccination against varicella.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Subjects with blood dyscrasias, leukemia, and lymphomas of any type.
* A family history of congenital or hereditary immunodeficiency
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including hypersensitivity to neomycin or latex.
* Major congenital defects or serious chronic illness.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥38. 0°C/100.4°F by any age appropriate route.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Active untreated tuberculosis based on medical history.
* Any other condition which, in the opinion of the investigator, prevents the child from participating in the study.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1236 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (12):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Schönau am Königssee, Bavaria
  - GSK Investigational Site, Vellmar, Hesse
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Wurzen, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Neumünster
- Mexico (2):
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Mexico City
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (4):
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19836

REFERENCES:
- [Background] Faust SN, Le Roy M, Pancharoen C, Weber MAR, Cathie K, Behre U, Bernatoniene J, Snape MD, Helm K, Medina Pech CE, Henry O, Baccarini C, Povey M, Gillard P. Safety and immunogenicity of a varicella vaccine without human serum albumin (HSA) versus a HSA-containing formulation administered in the second year of life: a phase III, double-blind, randomized study. BMC Pediatr. 2019 Feb 7;19(1):50. doi: 10.1186/s12887-019-1425-7. PMID 30732648

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five vaccinated subjects for whom the data could not be used due to invalid informed consent were excluded.
Groups:
- VAR_HSA_F Group: 2 doses of Varilrix HSA-free vaccine, one at Visit 1 (Day 0) and the other at Visit 2 (Day 42), were given to the subjects in this group. The vaccine was administered subcutaneously in the triceps region of the left arm
- VAR Group: 2 doses of Varilrix™ vaccine, one at Visit 1 (Day 0) and the other at Visit 2 (Day 42), were given to the subjects in this group. The vaccine was administered subcutaneously in the triceps region of the left arm
Period: Overall Study
Arm/Group | VAR_HSA_F Group | VAR Group
Started | 615 | 616
Completed | 609 | 607
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 2 | 0
Not completed — Unable To Arrange Visit 3 | 1 | 0
Not completed — Violation Of Procedures GSK | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAR_HSA_F Group | VAR Group | Total
Number analyzed (Participants) | 615 | 616 | 1231
Age, Continuous [Mean (Standard Deviation); unit: Months] | 16.7 (3.3) | 16.9 (3.4) | 16.8 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 318 | 312 | 630
  Male | 297 | 304 | 601
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 3 | 1 | 4
  Asian - Central/South Asian Heritage | 2 | 2 | 4
  Asian - East Asian Heritage | 3 | 2 | 5
  Asian - South East Asian Heritage | 133 | 135 | 268
  Other | 94 | 94 | 188
  White - Arabic / North African Heritage | 1 | 1 | 2
  White - Caucasian / European Heritage | 379 | 381 | 760

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Fever
Description: Fever was defined as axillary temperature above (>) 39.0 °C (> 102.2°F)
Time Frame: 15-days (Days 0-14) post Dose 1 of varicella vaccination
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects with administration of either Varilrix HSA-free or Varilrix™vaccine documented. Number of participants analysed corresponds to the subjects in the Total Vaccinated cohort with documented dose 15-days (Days 0-14) post Dose 1 of varicella vaccination
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 612 | 614
Subjects | 24 | 32
Statistical Analysis 1: Comparison: VAR_HSA_F Group vs VAR Group; Non-inferiority of Varilrix HSA-free vaccine to Varilrix™ vaccine in terms of percentage of subjects reporting fever > 39.0°C (> 102.2°F) within 15-days (Days 0-14) after Dose 1 (VAR_HSA_F Group minus VAR Group); Test type: Non-Inferiority — Criterion for the Varilrix HSA-free vaccine as compared to Varilrix™ vaccine, the upper limit (UL) of the 2-sided standardised asymptotic 95% confidence interval (CI) for the group difference (VAR_HSA_F minus VAR) in incidence of fever > 39.0°C (> 102.2°F) within 0-14 days after Dose 1 was to be equal to or below 5%; Difference in percentage between groups = -1.29, 95% CI 2-sided [-3.72 to 1.08] — Power obtained using PASS 2005 (Likelihood Score [Miettinen and Nurminen approach]), one-sided non-inferiority test for the difference of two independent proportions, under the alternative associated to the reference value & alpha=2.5%

2. Secondary Outcome: Number of Subjects Reporting Fever
Description: Fever was defined as axillary temperature greater than or equal to (≥) 38.0°C (≥ 100.4°F)
Time Frame: 15 days post each dose of varicella vaccination
Population: Analysis was performed on the Total Vaccinated cohort. Number of participants analysed corresponds to the subjects in the Total Vaccinated cohort with documented dose 15-days post each dose of varicella vaccination for each of the 2 groups (VAR_HSA_F Group and VAR Group)
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 612 | 614
Subjects
  Fever ≥ 38 °C following Dose 1 | 83 | 92
  Fever ≥ 38 °C following Dose 2: number analyzed (Participants) | 611 | 610
  Fever ≥ 38 °C following Dose 2 | 83 | 86

3. Secondary Outcome: Evaluation of Immune Response to Varicella Vaccine With Respect to Anti Varicella Zoster Virus (Anti-VZV) Antibody Concentrations (Immuno-sub Cohort)
Description: Anti-VZY antibody concentrations were expressed in terms of Geometric Mean Concentrations (GMCs)
Time Frame: At Day 42 and Day 84 post vaccination
Population: Immunogenicity analyses were performed on the According-to-protocol (ATP) cohort for immunogenicity. Immune response (in terms of GMC) was assessed in sub cohort of the ATP cohort for immunogenicity for each group (immuno sub cohort) who had blood taken and tested for anti-varicella antibodies at Day 0, Day 42, and Day 84
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 185 | 173
mIU/mL
  Post Dose 1 blood sample at Day 42: number analyzed (Participants) | 185 | 168
  Post Dose 1 blood sample at Day 42 | 139.9 [126.7 to 154.5] | 146.0 [132.5 to 160.7]
  Post Dose 2 blood sample at Day 84: number analyzed (Participants) | 180 | 173
  Post Dose 2 blood sample at Day 84 | 931.8 [841.1 to 1032.3] | 1102.4 [996.1 to 1220.2]

4. Secondary Outcome: Number of Subjects With a Seroresponse to VZV (Immuno Sub Cohort)
Description: For VZV, seroresponse was defined as, post-vaccination anti-VZV antibody concentration ≥ 50 mIU/mL among subjects who were seronegative (antibody concentration below (< ) 25 mIU/mL) before vaccination
Time Frame: At Day 42 and Day 84 post vaccination
Population: Immunogenicity analyses were performed on the According-to-protocol (ATP) cohort for immunogenicity. Seropositivity was assessed in sub cohort of the ATP cohort for immunogenicity for each group (immuno sub cohort) who had blood taken and tested for anti-varicella antibodies at Day 0, Day 42, and Day 84
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 185 | 173
Subjects
  ≥ 25 mIU/mL (At Day 42): number analyzed (Participants) | 185 | 168
  ≥ 25 mIU/mL (At Day 42) | 184 | 168
  ≥ 50 mIU/mL (At Day 42): number analyzed (Participants) | 185 | 168
  ≥ 50 mIU/mL (At Day 42) | 174 | 166
  ≥ 25 mIU/mL (At Day 84): number analyzed (Participants) | 180 | 173
  ≥ 25 mIU/mL (At Day 84) | 180 | 173
  ≥ 50 mIU/mL (At Day 84): number analyzed (Participants) | 180 | 173
  ≥ 50 mIU/mL (At Day 84) | 180 | 173

5. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, injection site redness and swelling. Any = occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain = subject crying when limb was moved or as spontaneously painful. Grade 3 redness and swelling = above (>) 20 mm
Time Frame: 4-day post vaccination period following Dose 1 (Day 0) and Dose 2 (Day 42)
Population: Analysis was performed on the Total Vaccinated cohort. Number of participants analysed corresponds to the subjects in the Total Vaccinated cohort with at least one documented dose 4 days following each vaccination and across doses for each of the 2 groups (VAR_HSA_F Group and VAR Group)
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 612 | 614
Subjects
  Any Pain, Dose 1: number analyzed (Participants) | 612 | 613
  Any Pain, Dose 1 | 75 | 86
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 612 | 613
  Grade 3 Pain, Dose 1 | 2 | 4
  Any Redness, Dose 1: number analyzed (Participants) | 612 | 613
  Any Redness, Dose 1 | 149 | 150
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 612 | 613
  Grade 3 Redness, Dose 1 | 3 | 2
  Any Swelling, Dose 1: number analyzed (Participants) | 612 | 613
  Any Swelling, Dose 1 | 43 | 42
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 612 | 613
  Grade 3 Swelling, Dose 1 | 2 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 610 | 610
  Any Pain, Dose 2 | 63 | 80
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 610 | 610
  Grade 3 Pain, Dose 2 | 1 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 610 | 610
  Any Redness, Dose 2 | 168 | 185
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 610 | 610
  Grade 3 Redness, Dose 2 | 10 | 8
  Any Swelling, Dose 2: number analyzed (Participants) | 610 | 610
  Any Swelling, Dose 2 | 69 | 71
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 610 | 610
  Grade 3 Swelling, Dose 2 | 1 | 4
  Any Pain, Across Doses | 101 | 126
  Grade 3 Pain, Across Doses | 3 | 5
  Any Redness, Across Doses | 224 | 234
  Grade 3 Redness, Across Doses | 13 | 10
  Any Swelling, Across Doses | 92 | 94
  Grade 3 Swelling, Across Doses | 3 | 4

6. Secondary Outcome: Number of Subjects Reporting Fever
Description: Any fever (≥ 38°C) = occurrence of any fever regardless of its intensity grade or relationship to vaccination. Grade 3 fever = temperature > 39.5°C. Related fever = assessed by the investigator as causally related to study vaccination
Time Frame: 43-day post vaccination period following Dose 1 (Day 0) and Dose 2 (Day 42)
Population: Analysis was performed on the Total Vaccinated cohort. Number of participants analysed corresponds to the subjects in the Total Vaccinated cohort with the documented dose 43 days following each vaccination and across doses for each of the 2 groups (VAR_HSA_F Group and VAR Group)
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 612 | 614
Subjects
  Fever (Axillary), Dose 1 : ≥ 38 °C | 205 | 188
  Fever (Axillary), Dose 1 : > 39.5 °C | 40 | 27
  Fever (Axillary), Dose 1 : Related | 72 | 51
  Fever (Axillary), Dose 2 : ≥ 38 °C: number analyzed (Participants) | 611 | 610
  Fever (Axillary), Dose 2 : ≥ 38 °C | 172 | 177
  Fever (Axillary), Dose 2 : > 39.5 °C: number analyzed (Participants) | 611 | 610
  Fever (Axillary), Dose 2 : > 39.5 °C | 23 | 31
  Fever (Axillary), Dose 2 : Related: number analyzed (Participants) | 611 | 610
  Fever (Axillary), Dose 2 : Related | 51 | 57
  Fever (Axillary), Across Doses : ≥ 38 °C | 301 | 290
  Fever (Axillary), Across Doses : > 39.5 °C | 57 | 53
  Fever (Axillary), Across Doses : Related | 111 | 95

7. Secondary Outcome: Number of Subjects Reporting Rash
Description: Any rash = occurrence of the specified solicited general symptom regardless of its intensity. Grade 3 rash = rash which prevented normal, everyday activities. Related rash = assessed by the investigator as causally related to study vaccination
Time Frame: 43-day post vaccination period following Dose 1 (Day 0) and Dose 2 (Day 42)
Population: Analysis was performed on the Total Vaccinated cohort. Number of participants analysed corresponds to the subjects in the Total Vaccinated cohort with at least one documented dose 43 days following each vaccination and across doses for each of the 2 groups (VAR_HSA_F Group and VAR Group)
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 612 | 614
Subjects
  Any, Dose 1 : Localised or generalised | 89 | 104
  Any, Dose 1 : With fever | 32 | 27
  Any, Dose 1 : Varicella like | 7 | 9
  Any, Dose 1 : Grade 3 | 2 | 4
  Any, Dose 1 : Related | 16 | 23
  Localised, Dose 1 : Any | 65 | 74
  Localised, Dose 1 : Administration site | 4 | 2
  Localised, Dose 1 : Other site | 63 | 72
  Localised, Dose 1 : With fever | 18 | 12
  Localised, Dose 1 : Varicella like | 5 | 4
  Localised, Dose 1 : Grade 3 | 2 | 1
  Localised, Dose 1 : Related | 11 | 13
  Generalised, Dose 1 : Any | 29 | 35
  Generalised, Dose 1 : With fever | 14 | 15
  Generalised, Dose 1 : Varicella like | 2 | 6
  Generalised, Dose 1 : Grade 3 | 0 | 3
  Generalised, Dose 1 : Related | 5 | 11
  Any, Dose 2 : Localised or generalised: number analyzed (Participants) | 611 | 610
  Any, Dose 2 : Localised or generalised | 76 | 78
  Any, Dose 2 : With fever: number analyzed (Participants) | 611 | 610
  Any, Dose 2 : With fever | 27 | 34
  Any, Dose 2 : Varicella like: number analyzed (Participants) | 611 | 610
  Any, Dose 2 : Varicella like | 4 | 5
  Any, Dose 2 : Grade 3: number analyzed (Participants) | 611 | 610
  Any, Dose 2 : Grade 3 | 2 | 5
  Any, Dose 2 : Related: number analyzed (Participants) | 611 | 610
  Any, Dose 2 : Related | 15 | 16
  Localised, Dose 2 : Any: number analyzed (Participants) | 611 | 610
  Localised, Dose 2 : Any | 52 | 57
  Localised, Dose 2 : Administration site: number analyzed (Participants) | 611 | 610
  Localised, Dose 2 : Administration site | 1 | 4
  Localised, Dose 2 : Other site: number analyzed (Participants) | 611 | 610
  Localised, Dose 2 : Other site | 51 | 53
  Localised, Dose 2 : With fever: number analyzed (Participants) | 611 | 610
  Localised, Dose 2 : With fever | 16 | 23
  Localised, Dose 2 : Varicella like: number analyzed (Participants) | 611 | 610
  Localised, Dose 2 : Varicella like | 3 | 2
  Localised, Dose 2 : Grade 3: number analyzed (Participants) | 611 | 610
  Localised, Dose 2 : Grade 3 | 1 | 1
  Localised, Dose 2 : Related: number analyzed (Participants) | 611 | 610
  Localised, Dose 2 : Related | 12 | 9
  Generalised, Dose 2 : Any: number analyzed (Participants) | 611 | 610
  Generalised, Dose 2 : Any | 25 | 26
  Generalised, Dose 2 : With fever: number analyzed (Participants) | 611 | 610
  Generalised, Dose 2 : With fever | 11 | 12
  Generalised, Dose 2 : Varicella like: number analyzed (Participants) | 611 | 610
  Generalised, Dose 2 : Varicella like | 1 | 3
  Generalised, Dose 2 : Grade 3: number analyzed (Participants) | 611 | 610
  Generalised, Dose 2 : Grade 3 | 1 | 4
  Generalised, Dose 2 : Related: number analyzed (Participants) | 611 | 610
  Generalised, Dose 2 : Related | 3 | 8
  Any, Across Doses : Localised or generalised | 144 | 152
  Any, Across Doses : With fever | 55 | 59
  Any, Across Doses : Varicella like | 11 | 14
  Any, Across Doses : Grade 3 | 4 | 9
  Any, Across Doses : Related | 28 | 37
  Localised, Across Doses : Any | 106 | 112
  Localised, Across Doses : Administration site | 5 | 6
  Localised, Across Doses : Other site | 103 | 107
  Localised, Across Doses : With fever | 32 | 34
  Localised, Across Doses : Varicella like | 8 | 6
  Localised, Across Doses : Grade 3 | 3 | 2
  Localised, Across Doses : Related | 20 | 21
  Generalised, Across Doses : Any | 49 | 57
  Generalised, Across Doses : With fever | 24 | 27
  Generalised, Across Doses : Varicella like | 3 | 9
  Generalised, Across Doses : Grade 3 | 1 | 7
  Generalised, Across Doses : Related | 8 | 19

8. Secondary Outcome: Number of Subjects Reporting Febrile Convulsions
Description: Any febrile convulsion = occurrence of the specified solicited general symptom regardless of its intensity. Grade 3 febrile convulsion = febrile convulsion which prevented normal, everyday activities. Related febrile convulsion = assessed by the investigator as causally related to study vaccination
Time Frame: 43-day post vaccination period following Dose 1 (Day 0) and Dose 2 (Day 42)
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 612 | 614
Subjects
  Febrile convulsion, Dose 1 : Any | 1 | 1
  Febrile convulsion, Dose 1 : Grade 3 | 0 | 1
  Febrile convulsion, Dose 1 : Related | 0 | 0
  Febrile convulsion, Dose 2 : Any: number analyzed (Participants) | 611 | 610
  Febrile convulsion, Dose 2 : Any | 0 | 1
  Febrile convulsion, Dose 2 : Grade 3: number analyzed (Participants) | 611 | 610
  Febrile convulsion, Dose 2 : Grade 3 | 0 | 0
  Febrile convulsion, Dose 2 : Related: number analyzed (Participants) | 611 | 610
  Febrile convulsion, Dose 2 : Related | 0 | 0
  Febrile convulsion, Across Doses : Any | 1 | 2
  Febrile convulsion, Across Doses : Grade 3 | 0 | 1
  Febrile convulsion, Across Doses : Related | 0 | 0

9. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination
Time Frame: 43-day post vaccination period following Dose 1 (Day 0) and Dose 2 (Day 42)
Population: Analysis was performed on the Total Vaccinated cohort. Number of participants analysed corresponds to the subjects in the Total Vaccinated cohort with the administered dose 43 days following each vaccination and across doses for each of the 2 groups (VAR_HSA_F Group and VAR Group)
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 615 | 616
Subjects
  Post Dose 1 | 270 | 282
  Post Dose 2: number analyzed (Participants) | 611 | 611
  Post Dose 2 | 223 | 220

10. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life threatening, required hospitalisation or prolongation of hospitalisation or resulted in disability/incapacity. Any SAE = occurrence of SAE regardless of intensity grade or relation to vaccination
Time Frame: From Day 0 through the end of study (Day 84)
Measure: Number; unit: Subjects
Arm/Group | VAR_HSA_F Group | VAR Group
Number analyzed (Participants) | 615 | 616
Subjects | 13 | 15

ADVERSE EVENTS:
Time Frame: Solicited local AEs: During the 4-day post vaccination period after each dose. Solicited general and unsolicited AEs: During the 43-day post vaccination period after each dose. Serious adverse events: From Day 0 through the end of study (Day 84)
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed
Arm/Group | VAR_HSA_F Group | VAR Group
All-Cause Mortality (participants affected / at risk) | 0/615 | 0/616
Serious Adverse Events (participants affected / at risk) | 13/615 | 15/616
Other Adverse Events (participants affected / at risk) | 489/615 | 491/616
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAR_HSA_F Group (N=615) | VAR Group (N=616)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (7) | 3 (3)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pseudocroup (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAR_HSA_F Group (N=615) | VAR Group (N=616)
Cough (Respiratory, thoracic and mediastinal disorders) | 57 (71) | 49 (59)
Diarrhoea (Gastrointestinal disorders) | 38 (44) | 39 (53)
Injection site erythema (General disorders) | 224 (319) | 237 (341)
Injection site pain (General disorders) | 101 (138) | 127 (167)
Injection site swelling (General disorders) | 92 (112) | 95 (114)
Nasopharyngitis (Infections and infestations) | 87 (110) | 80 (102)
Pyrexia (General disorders) | 301 (377) | 290 (365)
Rash (Skin and subcutaneous tissue disorders) | 144 (165) | 152 (182)
Rhinitis (Infections and infestations) | 33 (40) | 25 (32)
Teething (Gastrointestinal disorders) | 58 (130) | 55 (80)
Upper respiratory tract infection (Infections and infestations) | 28 (35) | 37 (42)
Vomiting (Gastrointestinal disorders) | 31 (34) | 34 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.